CLINICAL TRIAL: NCT01084070
Title: Randomized Clinical Trial of Early Oral Feeding Versus Traditional Postoperative Care in Emergency Abdominal Surgery
Brief Title: Early Oral Feeding Versus Traditional Postoperative Care in Emergency Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General de Agudos "Dr. Cosme Argerich" (Other)
Responsible Party: Principal Investigator, Klappenbach Roberto, Investigator, Hospital General de Agudos "Dr. Cosme Argerich"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ARGERICH1
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Postoperative Care
Keywords: early feeding; postoperative care; emergency surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early oral feeding (Experimental)
  Interventions: Other: Early oral feeding
- Traditional Care (Active Comparator)
  Interventions: Other: Traditional Care

INTERVENTIONS:
Other: Early oral feeding — Within 6-24 hours after surgery the nasogastric tube will be removed and liquids and soft diet "at will" indicated.
  Arms: Early oral feeding
Other: Traditional Care — They will have nasogastric tube and restriction of oral intake until the first sign of restoration of intestinal transit (first flatus or stool, whichever comes first). Since then withdrew nasogastric tube and liquid diet starts within 24 hours, then continues with soft diet.
  Arms: Traditional Care

SUMMARY:
The traditional postoperative care after abdominal surgery included the need of nasogastric tube, fasting until resumed bowel function and progressive reinstitution of oral intake from liquid to solid diet. Recent studies have shown no benefits of this traditional management over early oral feeding. Nevertheless, the researches in emergency surgery are scarce.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14 years after abdominal emergency surgery.

Exclusion Criteria:

* Lack of consensus of the patient
* Concurrent extra-abdominal surgery
* Short bowel or other clear indication of parenteral nutrition
* Inability to feed orally (eg, decreased level of consciousness)
* Interventional procedure
* Esophageal surgery
* Reoperations
* Pancreatitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | At 30 days or at discharge
  The rate of postoperative complications according with Clavien-Dindo classification, defined as "any deviation from the normal postoperative course".

SECONDARY OUTCOMES:
Gastrointestinal leaks | At 30 days or at discharge
  "the leak of luminal contents from a surgical join between two hollow viscera or from surgical repair of continuity solution. The luminal contents may emerge either through the wound or at the drain site, or they may collect near the anastomosis or rapair, causing fever, abscess, septicaemia, metabolic disturbance and/or multiple-organ failure. The escape of luminal contents intoan adjacent localised area, detected by imaging, in the absence of clinical symptoms and signs should be recorded as a subclinical leak"
Time to resume bowel functions | At 30 days or at discharge
  Time from surgery to the first flatus or deposition, whatever occurs first
Oral diet intolerance | At 30 days or at discharge
  The appearance of vomits or abdominal pain after diet
Postoperative hospital stay | At 90 days
  Postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Klappenbach, MD, Principal Investigator — Argerich Hospital
Locations (1):
- Argerich Hospital, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Klappenbach RF, Yazyi FJ, Alonso Quintas F, Horna ME, Alvarez Rodriguez J, Oria A. Early oral feeding versus traditional postoperative care after abdominal emergency surgery: a randomized controlled trial. World J Surg. 2013 Oct;37(10):2293-9. doi: 10.1007/s00268-013-2143-1. PMID 23807124